CLINICAL TRIAL: NCT02427035
Title: A Double-blind, Randomized, Placebo-controlled, Pharmacokinetic, Safety and Tolerability Study of CSL112 in Adult Subjects With Moderate Renal Impairment and in Healthy Adult Subjects With Normal Renal Function
Brief Title: A Study of CSL112 in Healthy Adults and in Adults With Moderate Renal Impairment
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: CSL Behring (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CSL112_1001; 2014-005520-10 (EudraCT Number)
Record Dates: First submitted 2015-04-20; First posted 2015-04-27 (Estimated); Last update posted 2017-09-19 (Actual); Status verified 2017-09

CONDITIONS: Acute Myocardial Infarction
MeSH Terms: interventions — CSL112

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Low (Experimental): A low dose of either CSL112 or placebo is to be administered as a single intravenous (IV) infusion. The placebo will be administered at the same frequency, volume and duration as the CSL112 infusion.
  Interventions: Biological: CSL112; Other: Placebo
- High (Experimental): A high dose of either CSL112 or placebo is to be administered as a single intravenous (IV) infusion. The placebo will be administered at the same frequency, volume and duration as the CSL112 infusion.
  Interventions: Biological: CSL112; Other: Placebo

INTERVENTIONS:
Biological: CSL112 — CSL112 is a novel formulation of apolipoprotein A-I (apoA-I) purified from human plasma and reconstituted to form high-density lipoprotein (HDL) particles.
Other: Placebo — 0.9% weight/volume sodium chloride solution (ie, normal saline)

SUMMARY:
This is a phase 1 multicenter, randomized, double-blind, placebo-controlled, ascending dose study to investigate the pharmacokinetics (PK), safety, and tolerability of CSL112 in adult subjects with moderate renal impairment and in healthy adult subjects with normal renal function.

ELIGIBILITY:
Inclusion Criteria:

* Men or women aged 18 to 85 years (inclusive) of age, with body weight 50 kg or more.
* Subjects with renal impairment (RI) must have stable chronic moderate RI (estimated glomerular filtration rate [eGFR] ≥ 30 and < 60 mL/min/1.73 m2)
* Healthy subjects must have normal renal function (eGFR ≥ 90 mL/min/1.73 m2)

Exclusion Criteria:

* Evidence of a clinically significant medical condition, disorder or disease
* Evidence of hepatobiliary disease
* Any clinically relevant abnormal laboratory test result
* Known history of allergies, hypersensitivity or deficiencies to CSL112 or any of its components
* Other severe comorbid condition, concurrent medication, or other issue that renders the subject unsuitable for participation in the study, including: history of cancer, low platelet count, bleeding disorder or coagulopathy, significantly altered electrocardiogram waveform, unstable glycemia control in subjects with diabetes, acute renal failure, recent donation or loss of blood
* Evidence or history of alcohol or substance abuse

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2015-05; Primary Completion 2015-11 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Plasma apolipoprotein A-I (apoA-I) and phosphatidylcholine (PC) area under the curve (AUC) | Before and at up to 10 time points (during up to 7 days) after infusion
  Baseline corrected plasma apoA-I and PC AUC0-infinity
Plasma apoA-I and PC AUC0-last and AUC 0-t | Before and at up to 10 time points (during up to 7 days) after infusion
  AUC from time point zero to the last quantifiable time point before the analyte first returns to baseline (AUC0-last) and/or a partial AUC from baseline to time point t (AUC0-t) with and without baseline correction
Plasma apoA-I and PC Cmax | Before and at up to 10 time points (during up to 7 days) after infusion
Plasma apoA-I and PC Tmax | Before and at up to 10 time points (during up to 7 days) after infusion
Plasma apoA-I and PC Volume of distribution during terminal phase | Before and at up to 10 time points (during up to 7 days) after infusion
Plasma apoA-I and PC clearance | Before and at up to 10 time points (during up to 7 days) after infusion
Plasma apoA-I and PC t1/2 | Before and at up to 10 time points (during up to 7 days) after infusion
Urinary excretion of apoA-I (Ae0-t) | Before and up to 48 hours after infusion
  Amount excreted (Ae) of apoA-I over a collection interval 0-t.
Urinary excretion of apoA-I (%fe0-t) | Before and up to 48 hours after infusion
  Percent fraction excreted (%fe) of apoA-I in urine over time interval 0-t, calculated as Ae0-t/Dose x 100.
Renal clearance of apoA-I | Before and up to 48 hours after infusion
  Renal clearance of apoA-I, calculated as Ae0-48/AUC0-48

SECONDARY OUTCOMES:
Urinary excretion of sucrose(Ae0-t) | Before and up to 48 hours after infusion
  Amount of sucrose excreted over a collection interval 0-t.
Urinary excretion of sucrose (%fe0-t) | Before and up to 48 hours after infusion
  Percent fraction excreted sucrose in urine over time interval 0-t, calculated as Ae0-t/Dose x 100.
Urinary excretion of sucrose (clearance) | Before and up to 48 hours after infusion
  Renal clearance of sucrose, calculated as Ae0-48/AUC0-48
Adverse drug reaction (ADR) or suspected ADR frequency (%) | Up to approximately 127 days
  The overall percentage of participants with adverse reactions or suspected adverse reactions:
  1. That begin during or within 1 hour of an infusion; or
  2. That may be causally related to the administration of the investigational product; or
  3. For which the Investigator's causality assessment is missing or indeterminate; or
  4. For which the incidence in an active treatment arm exceeds the exposure-adjusted incidence rate in the placebo arm by 30% or more, provided the difference in incidence rates is 1% or more.
Clinically significant changes in routine safety assessments | Up to approximately 97 days
  The number of participants with clinically significant changes in any of the following assessments: clinical laboratory tests, physical examinations, body weight, electrocardiograms, vital signs, immunogenicity testing, serology, nucleic acid testing or proteinuria findings.
Clinically important change in drug-induced liver injury | From baseline (before infusion) up to Day 16.
  A clinically important change in drug-induced liver injury is defined as a change (from baseline) in alanine aminotransferase (ALT) greater than 3 times the upper limit of normal (ULN) or a change in total bilirubin greater than 2 times ULN, that is confirmed upon repeat measurement.
Clinically important change in renal status | From baseline (before infusion) up to Day 16.
  A clinically important change in renal status is defined as a serum creatinine (Cr) increase to ≥ 1.5 x the baseline value that is confirmed upon repeat measurement, or the need for renal replacement therapy.
Plasma sucrose AUC | Before and at up to 7 time points (during up to 2 days) after infusion
  Baseline corrected plasma sucrose AUC0-infinity
Plasma sucrose AUC0-last and AUC 0-t | Before and at up to 7 time points (during up to 2 days) after infusion
  AUC from time point zero to the last quantifiable time point before the analyte first returns to baseline (AUC0-last) and/or a partial AUC from baseline to time point y (AUC0-t) with and without baseline correction
Plasma sucrose Cmax | Before and at up to 7 time points (during up to 2 days) after infusion
Plasma sucrose Tmax | Before and at up to 7 time points (during up to 2 days) after infusion
Plasma sucrose Volume of distribution during terminal phase | Before and at up to 7 time points (during up to 2 days) after infusion
Plasma sucrose Clearance | Before and at up to 7 time points (during up to 2 days) after infusion
Plasma sucrose t1/2 | Before and at up to 7 time points (during up to 2 days) after infusion
Adverse drug reaction (ADR) or suspected ADR frequency | Up to approximately 127 days
  The overall number of participants with adverse reactions or suspected adverse reactions:
  1. That begin during or within 1 hour of an infusion; or
  2. That may be causally related to the administration of the investigational product; or
  3. For which the Investigator's causality assessment is missing or indeterminate; or
  4. For which the incidence in an active treatment arm exceeds the exposure-adjusted incidence rate in the placebo arm by 30% or more, provided the difference in incidence rates is 1% or more.
Number of subjects with AEs | After the start of infusion up to approximately 127 days

CONTACTS AND LOCATIONS:
Overall Officials: Denise D'Andrea, M.D., Study Director — CSL Behring
Locations (4):
- Germany (2):
  - Study Site - 17101, Berlin
  - Study Site - 17102, Munich
- United Kingdom (2):
  - Study Site - 24101, London
  - Study Site - 24102, Manchester

REFERENCES:
- [Derived] Zheng B, Duffy D, Tricoci P, Kastrissios H, Pfister M, Wright SD, Gille A, Tortorici MA. Pharmacometric analyses to characterize the effect of CSL112 on apolipoprotein A-I and cholesterol efflux capacity in acute myocardial infarction patients. Br J Clin Pharmacol. 2021 Jun;87(6):2558-2571. doi: 10.1111/bcp.14666. Epub 2020 Dec 23. PMID 33217027
- [Derived] Tortorici MA, Duffy D, Evans R, Feaster J, Gille A, Mant TGK, Wright SD, D'Andrea D. Pharmacokinetics and Safety of CSL112 (Apolipoprotein A-I [Human]) in Adults With Moderate Renal Impairment and Normal Renal Function. Clin Pharmacol Drug Dev. 2019 Jul;8(5):628-636. doi: 10.1002/cpdd.618. Epub 2018 Sep 21. PMID 30240132